CLINICAL TRIAL: NCT05684926
Title: Investigation of the Effect of Yoga Training With Telerehabilitation on Asthma Control, Functional Capacity, Physical Fitness, Physical Activity and Quality of Life in Children With Asthma During the COVID-19 Pandemic Process
Brief Title: COVID-19 Pandemic Asthma Child Telerehabilitation Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Şeyma Nur Önal, Lecturer, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA22030
Record Dates: First submitted 2023-01-12; First posted 2023-01-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Asthma in Children; Telerehabilitation; Yoga
Keywords: Asthma; Rehabilitation; Physical Fitness; Physical activity
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The intervention group is a group of asthmatic children aged 6-11 years, determined by randomization. Yoga asana includes pranayama and concentration. It will be held 3 days a week for 12 weeks.
  Interventions: Other: Telerehabilitation yoga
- Control Group (No Intervention): The control group is a group of asthmatic children aged 6-11 years, determined by randomization method. He will be put on the waiting list and after the second evaluation, yoga exercises will be done for 8 weeks.

INTERVENTIONS:
Other: Telerehabilitation yoga — Yoga consists of bodily postures or poses called asanas, breathing practices called pranayama, and meditation sections that provide focus. Children's yoga aims to teach pre-school (3-6 years) and school (7-12 years) children to breathe correctly, to practice yoga postures using their imaginations, to preserve their existing body flexibility and to teach correct posture. It consists of compositions such as postures, breathing exercises, imitations of living things in nature, memory games. They also relax with the pranayama breathing exercises done during the session. It aims to develop children's creativity through relaxation exercises, moving poses and stories told. Children's yoga also serves an artistic aspect with activities such as listening to music, singing, rhythm games, and drawing.
  Other Names: Yoga/Pranayama
  Arms: Experimental Group

SUMMARY:
In our study, yoga asana and pranayama practices, which will be applied by video call from computer or phone, will be advantageous in terms of time, transportation and access to asthmatic children whose anxiety and anxiety levels increase during the COVID-19 period, whose access to hospital services is difficult, and whose physical activity level decreases due to the increase in screen time. It was aimed to examine the effects of these group exercises on Asthma Control, Functional Capacity, Physical Fitness, Physical Activity and Quality of Life. In the randomized controlled study, the treatment and control group will be determined by the closed envelope method, the control group will be placed on the waiting list and yoga will be practiced at the end of the study. The first and final evaluation will be done face to face in a clinical setting. The total duration will be 12 weeks, 3 days a week and 36 sessions between 8-8:40 in the evening. Researchers who will do yoga have a certificate of practice. Patients will be followed up in Hacettepe University Medical Faculty Asthma Allergy Clinic.

DETAILED DESCRIPTION:
In our study, yoga asana and pranayama practices, which will be applied by video call from computer or phone, will be advantageous in terms of time, transportation and access to asthmatic children whose anxiety and anxiety levels increase during the COVID-19 period, whose access to hospital services is difficult, and whose physical activity level decreases due to the increase in screen time. It was aimed to examine the effects of these group exercises on Asthma Control, Functional Capacity, Physical Fitness, Physical Activity and Quality of Life. In the randomized controlled study, the treatment and control group will be determined by the closed envelope method, the control group will be placed on the waiting list and yoga will be practiced at the end of the study. The first and final evaluation will be done face to face in a clinical setting. Researchers who will do yoga have a certificate of practice. Patients will be followed up in Hacettepe University Medical Faculty Asthma Allergy Clinic. At the end of the study, pulmonary function assessment will be made for primary outcomes. Asthma control, functional testing, and quality of life will be evaluated for secondary outcomes. This study consists of a total of 36 sessions, 3 sessions per week for 12 weeks, and sessions of 40-50 minutes, and the measurements of these values at the beginning and after 36 sessions will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Hacettepe University Faculty of Medicine, Department of Pediatrics, Allergy and Asthma Unit patients were referred for Cardiopulmonary Rehabilitation,
* Those who have been diagnosed with asthma,
* Not in an asthma attack but clinically stable,
* Between the ages of 6-11,
* Giving consent on a voluntary basis,
* cooperative,
* Ability to use a smart phone or computer,

Exclusion Criteria:

* Individuals with internet connection will be included in the research. Individuals with asthma were included in the study.
* In an asthma attack and clinically unstable,
* Having serious diseases such as cancers, heart failure and acute respiratory infections,
* Having chronic lung disease other than asthma,
* Severe neuromuscular and musculoskeletal problems,
* Uncooperative to make surveys and scales,
* Admitted or hospitalized due to an asthma attack in the last 3 months for safety reasons,
* Having neuropsychiatric diseases,
* Individuals who do not volunteer to participate in the study will not be included in the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
respiratory function (pulmoner function test) | one day
  It is evaluated with the Pulmonary Function Test. After a deep, full inspiration, a forced expiratory maneuver is performed. Used with disposable antiviral filter. The patient's height and body weight are measured and recorded with age. It is done 3 times, there should be no more than 10% difference between the values. The highest value is accepted.

SECONDARY OUTCOMES:
asthma control | one day
  The Child Asthma Control Test (C-AKT) has a total of 7 items and covers the last 4 weeks. The first of the two sections is filled in by the child and consists of four questions about perception of asthma control, restriction of activities, coughing, and night awakenings. The second part is filled in by the parent or caregiver and consists of three questions (daytime complaints, daytime wheezing and night waking). The overall score ranges from 0 (poorest asthma control) to 27 (optimal asthma control).
functional capacity | one day
  six munite walk test It will be measured with the 6 Minute Walk Test. You can walk for 6 minutes at a fast pace without running in the 30 m long corridor. The distance walked is recorded. Vital values are recorded before and after.
physical fitness | one day
  FITNESSGRAM test batary The fitnessgram will be evaluated with the test battery. Valid from 5 years old. (a) Sit and lie down with back support (b) Trunk Extension (c) Trunk Lateral Flexion, Curl (d) Do push-ups. (e) For progressive aerobic cardiovascular endurance running (PACER), the time set for reaching 20 meters is 9 seconds, reduced by half a second per minute. If the rhythm cannot be kept up or the boundary line is not reached before the beep twice, the test is stopped and the number of laps is recorded.
physical activity | one day
  physical activity questionnaire child It examines the physical activity of children in the last seven days and the frequency of activities. It consists of 10 questions and a 5-point Likert structure. The first question questions activity and frequency. The 9th question questions the activity frequency on the days of the week. The remaining 8 questions evaluate sports, dance and play activity during the day or at certain time intervals throughout the week. Each question has a score of 1-5. The minimum score that can be obtained from the FAS is 9 and the maximum score is 45. The 10th question of the FAS questions any reason that prevents physical activity and is not scored.
pediatric asthma quality of life questionnaire | one day
  pediatric asthma quality of life questionnaire It was developed to measure the physical, mental and social disorders of children with asthma (7-17 years old). The scale, which questions the asthma experience in the last week, consists of 3 sub-units, namely 'symptoms', 'activity limitation' and 'emotional function', and 23 questions. Each question is in 7-point Likert type, showing 1- the worst and 7- the best situation. The score to be taken from the scale is between 23-167 and the total score is divided by the number of questions and scoring is done. A high score indicates good quality of life.
pediatric reach test | one day
  Evaluates the dynamic component of balance. It is performed by recording the distance in cm with a tape measure that they can reach forward and then to the right and left, respectively, without raising their heels from the ground in standing upright positions.
periferic muscle test | one day
  Peripheral Muscle Strength Hand Grip Test: Jamar hand dynamometer is used. The person sits in an upright position with the knees at 90°, the wrists are in neutral, the elbow is 90° and the dynamometer is gripped with all his strength, and the measurements are repeated 3 times on the right and left, with 10 seconds intervals.
  Quadriceps Muscle Strength: A hand-held dynamometer (Lafayette Manual Muscle Testing System; Lafayette Instrument Company, Lafayette, Indiana, USA) is used to measure lower extremity muscle strength. People sit with their knees and hips 90º. It is requested to maintain knee extension.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No